CLINICAL TRIAL: NCT05386706
Title: Treating Polycystic Ovarian Syndrome (PCOS) With Digital Intervention vs. Metformin
Brief Title: Treating PCOS With Digital Intervention vs. Metformin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Director, Principal Investigator, Clinical Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Digital Intervention PCOS
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Intervention (Experimental): A mini program-based digital intervention.
  Interventions: Behavioral: Digital Intervention
- Metformin (Active Comparator): Traditional metformin monotherapy.
  Interventions: Drug: Metformin

INTERVENTIONS:
Behavioral: Digital Intervention — This study developed a mini-program that combined diet, exercise, sleep, and mood interventions for PCOS women.
  Arms: Digital Intervention
Drug: Metformin — Traditional metformin monotherapy.
  Other Names: Metformin treatment
  Arms: Metformin

SUMMARY:
With the change in environment and lifestyle, and the improvement of people's understanding of PCOS, the incidence of PCOS is increasing worldwide. According to statistics, the prevalence of PCOS in premenopausal women is as high as 5-20%. Lifestyle interventions are the main treatment option for patients with PCOS. In addition, research has shown that digital therapy can effectively improve behavior changes in diet, exercise, and medication adherence, predict disease progression, reduce the frequency of disease-related symptoms, and promote effective disease management. This study aimed to investigate the efficacy of digital intervention versus traditional metformin monotherapy in patients with PCOS.

DETAILED DESCRIPTION:
This study developed a mini-program that combined diet, exercise, sleep, and mood interventions for PCOS women.

ELIGIBILITY:
Inclusion Criteria:

Female aged 18- 45; Meet Rotterdam criteria; Insulin Resistance

Exclusion Criteria:

Women who are pregnant or have a pregnancy plan within six months; Congenital adrenocortical hyperplasia; Hyperprolactinemia; Hyperthyroidism or hypothyroidism; Abnormal liver function (≥ 3 times the upper limit of the normal range); Abnormal renal function (GFR<60ml/min/1.73m2); Adrenal or ovarian tumors secreting androgens; Used contraceptives, metformin, pioglitazone, and antidepressant medication in the last 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Homeostasis model assessment of insulin resistance | 3 months
  insulin resistance index

SECONDARY OUTCOMES:
Anthropometry | 3 months
  body mass index (kg/m2)
menstrual frequency | 3 months
  number of menstruation in a year
fasting glucose | 3 months
  fasting glucose（mmol/L)
fasting insulin | 3 months
  fasting insulin（mmol/L)
Total cholesterol | 3 months
  Total cholesterol (mmol/L)
Triglycerides | 3 months
  Triglycerides (mmol/L)
HDL-c | 3 months
  HDL-c (mmol/L)
LDL-c | 3 months
  LDL-c (mmol/L)
total testosterone | 3 months
  total testosterone (nmol/L)
free testosterone | 3 months
  free testosterone (nmol/L)
Sex hormone-binding globulin | 3 months
  Sex hormone-binding globulin (nmol/L)
Androstenedione | 3 months
  Androstenedione (ng/ml)
Dehydroepiandrosterone | 3 months
  Dehydroepiandrosterone (ug/dl)
International Physical Activity Questionnaire (IPAQ) | 3 months
  Assess physical activity situation in women with PCOS.
Pittsburgh Sleep Quality Index (PSQI) | 3 months
  Assess sleep situation in women with PCOS.
Hospital Anxiety and Depression Scale (HADS) | 3 months
  To evaluate anxiety and depression in PCOS women.
Three-Factor Eating Questionnaire (TFEQ-R21) | 3 months
  Assess eating behavior in women with PCOS.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Doctor, Study Chair — Shanghai 10th People's Hospital
Locations (1):
- Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dilimulati D, Shao X, Wang L, Cai M, Zhang Y, Lu J, Wang Y, Liu H, Kuang M, Chen H, Zhang M, Qu S. Efficacy of WeChat-Based Digital Intervention Versus Metformin in Women With Polycystic Ovary Syndrome: Randomized Controlled Trial. J Med Internet Res. 2024 Oct 2;26:e55883. doi: 10.2196/55883. PMID 39357046